CLINICAL TRIAL: NCT07309861
Title: Effect Of Education On Adherence, Self Care And Well-Being Of Patients With Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Lale Yacan, Assistant Professor, Trakya University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TUTF-BAEK 2019/206
Record Dates: First submitted 2025-11-14; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease (Stage 3-4)
Keywords: Adaptation to illness; chronic kidney disease; self-care; well-being
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: The study population comprised of patients diagnosed with chronic kidney disease and receiving treatment in the nephrology outpatient clinic of a hospital. Considering the sample size of the study, since there are not sufficient data in the literature on the effect of the education provided to individuals with chronic kidney disease on adherence to illness, self-care, and well-being, it was calculated that 64 individuals from each group (intervention=64, control=64) should be included in the research with a power value of 80% and a margin of error of 5% to test the prediction of a medium effect size (d=0.5) of the education to be provided. Considering the possible losses during the study process, 70 individuals were included in each group.
  Patients were assigned to the intervention and control groups using the computer program Researcher Randomizer and the simple randomization method. In randomization between groups, characteristics such as age and sex of the patients who volunteered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effect of education on adherence, self care and well-being of patients with chronic kidney disease (Experimental): Patients who diagnosed with stage 3 to stage 4 chronic kidney disease
  Interventions: Device: Educational with chronic kidney disease

INTERVENTIONS:
Device: Educational with chronic kidney disease — Education Booklet for Patients with Chronic Kidney Disease It was prepared by the researchers in line with the literature review to be used as educational material for patients with stage 3 and stage 4 chronic kidney disease. The education booklet includes information about the kidneys (anatomy and functions of the kidneys), chronic kidney disease (definition of chronic kidney disease , risk factors, symptoms, nutrition in chronic kidney disease , salt consumption, the importance of potassium and phosphorus for our body, regular and balanced nutrition, exercise, the relationship between chronic kidney disease and diabetes, and the relationship between chronic kidney disease and hypertension), and treatment methods (hemodialysis, peritoneal dialysis, and kidney transplant).

SUMMARY:
ABSTRACT Aim: The aim of the study was evaluate the effect of education provided to patients diagnosed with chronic kidney disease on adherence to illness, self-care, and well-being.

Design: A randomised controlled trial. Participants: The study sample consisted of total of 119 individuals diagnosed with stage 3 to stage 4 chronic kidney disease.

Methods: The data were collected with the Patient Information Form, Adaptation to Chronic Illness Scale, Self-Care Management Process in Chronic Illness and the World Health Organization-5 Well-Being Index. The data were evaluated using descriptive analyses, the Mann-Whitney U test, Pearson's chi-square test, Fisher-Freeman test, student's t-test, Wilcoxon test, and Friedman test.

DETAILED DESCRIPTION:
Implications for the profession or patient care: This study contributes to the improvement of disease adaptation and self-care of individuals with stage 3 and stage chronic kidney disease.

Reporting Method: Consolidated Standards of Reporting Trials (CONSORT) Patient or Public Contribution: The study sample consisted of total of 119 individuals diagnosed with stage 3 to stage 4 chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* being over 18 years of age
* having stage 3 or stage 4 chronic kidney disease
* not having communication difficulties
* receiving outpatient treatment at the nephrology outpatient clinic
* and volunteering to take part in the research

Exclusion Criteria:

* being under 18 years of age
* having stage 1, 2 or stage 5 chronic kidney disease
* having communication difficulties
* not volunteering to take part in the research
* receiving hemodialysis or peritoneal dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Adaptation to Chronic Illness Scale | through study completion, an average of 19 months
  Adaptation to Chronic Illness Scale (ACIS): The scale includes 25 items, and a total score of 125 points is obtained from the scale. An increase in the scores from the subscales and/or the overall scale means that patients' adaptation levels to illness also increase.
The Self-Care Management Process in Chronic Illness (SCMP-G) | through study completion, an average of 19 months
  The Self-Care Management Process in Chronic Illness (SCMP-G): The scale includes 35 items and is evaluated as 5 (Strongly Agree) and 1 (Strongly Disagree). Self-care management increases with the increasing score on the scale.
WHO-5 Well-Being Index | through study completion, an average of 19 months
  WHO-5 Well-Being Index: The raw score is computed by summing the numbers belonging to 5 answers. Zero represents the worst possible quality of life, while 25 represents the best possible quality of life. To acquire a percentage score ranging from 0 to 100, the raw score is multiplied by 4. Whereas "zero percent" indicates the worst possible quality of life, "one hundred percent" indicates the best possible quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Özgül Erol, Professor, Study Director — Trakya University; Lale Yacan, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No